CLINICAL TRIAL: NCT01296139
Title: Evaluation of Ferumoxytol Enhanced MRI for the Detection of Lymph Node Involvement in Prostate Cancer
Brief Title: Ferumoxytol Enhanced MRI for the Detection of Lymph Node Involvement in Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 110098; 11-C-0098
Record Dates: First submitted 2011-02-12; First posted 2011-02-15 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2015-03-19

CONDITIONS: Prostate Cancer
Keywords: Non-Cutaneous Malignancy; Prostatectomy; Metastatic Prostate Cancer; Imaging Study; Magnetic Resonance Imaging; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ferrosoferric Oxide

ARMS (1):
- A (Experimental): All subjects will receive 7.5 mg/kg Fe
  Interventions: Drug: Ferumoxytol

INTERVENTIONS:
Drug: Ferumoxytol — All subjects will undergo pre-injection, 24, 48 hours post-Ferumoxytol injection (dose of 7.5mg/kg Fe) MRI consisting of T1 weighted (W), T2W and T2*W MRI in a 3 Tesla magnet. Additionally, all subjects will undergo pre-injection, 24 hours, 48 hours post-Ferumoxytol injection (dose of 7.5mg/kg Fe) ultrasound.

SUMMARY:
Background:

- Ferumoxytol is an approved iron replacement therapy agent that has some potential for use as a contrast agent in imaging studies of the lymph system, especially involving lymph nodes that have been affected by cancer. Ferumoxytol is taken up by normal lymph nodes, but excluded from cancerous lymph node tissue. Because Ferumoxytol has not yet been approved for use as an imaging agent, researchers are interested in testing its effectiveness as a contrast agent for studies of normal lymph tissue and cancer tissue in lymph nodes of individuals with prostate cancer.

Objectives:

- To evaluate the safety and effectiveness of Ferumoxytol as a contrast agent in individuals who are scheduled to have prostate removal surgery to treat prostate cancer.

Eligibility:

- Men at least 18 years of age who have been diagnosed with prostate cancer and are scheduled to have surgery to remove the prostate and surrounding lymph nodes.

Design:

* Participants will be screened with a full medical history and physical examination, blood and urine tests, and tumor imaging studies.
* Participants will have a magnetic resonance imaging (MRI) scan to provide baseline images for the study.
* Participants will receive an injection of Ferumoxytol and will return for another MRI scan on the following day (around 24 hours later).
* Some participants may have a third MRI scan 48 hours after the initial injection of Ferumoxytol. This third MRI scan is optional and not required by the study.
* Although the scanning and followup portion of the study will last only a few days, participants will be considered to be enrolled on the study until after the prostate removal surgery.

DETAILED DESCRIPTION:
Background:

* Prostate cancer is the most common non-cutaneous malignancy among men in Western world. Accurate lymph node staging is important in treatment planning for prostate cancer.
* Conventional imaging modalities (e.g. computed tomography [CT] and magnetic resonance imaging [MRI]) are used for the evaluation of lymph node involvement in many cancer types, including prostate cancer, however diagnosis is based on node enlargement which is neither sensitive nor specific in prostate cancer.
* As a consequence, the standard of care is to remove numerous lymph nodes during prostatectomy to ascertain lymph node status.
* A prior imaging agent for detecting lymph node involvement, dextran coated ultrasmall superparamagnetic iron oxide particles (USPIO), also known as Ferumoxtran-10 (Combidex , AMAG Pharmaceuticals, Inc. Lexington, MA, US) was shown to localize lymph node metastases with much greater accuracy than unenhanced MRI. Although a large study in lymph node imaging in prostate cancer was successfully conducted using ferumoxtran-10, the FDA Advisory Panel did not recommend broad use approval of this agent.
* A derivative of ferumoxtran-10, Ferumoxytol (Feraheme AMAG Pharmaceuticals, Inc. Lexington, MA, US) has been approved for iron replacement therapy. It is a semisynthetic carbohydrate coated, magnetic iron oxide preparation. This compound is taken up by normal lymph nodes, excluded from malignant nodal tissue. A single study of Ferumoxytol enhanced MRI demonstrated some efficacy of this agent at 24 hours but only one dose was used, MRI at later time points was not performed.
* Initial results of the NCI trial (11-C-0098) revealed that using the dose of 7.5 mg/kg Fe is safe and it yields a more homogenous and accurate signal changes in benign lymph nodes in comparison with the 4 and 6 mg/kg Fe doses. However, utility of this initial result could not be validated in depiction of signal change difference between benign and malignant lymph nodes with prostate cancer metastases.

Primary Objective

-To determine the optimal dose of Ferumoxytol for enhancing lymph nodes in patients with prostate cancer.

Eligibility

* Subject must be male and be (Bullet)18 years old.
* Subject must have a documented diagnosis of prostate cancer.

  --Those enrolling in the lymph node involvement subgroup must have imaging evidence of lymph node involvement (with a size of greater than or equal to 1.5cm)
* Eastern Cooperative Oncology Group Performance score of 0 to 2.
* Subjects must be scheduled to undergo prostatectomy and nodal dissection for presumed prostate cancer.

Design:

* Subjects with prostate cancer scheduled for prostatectomy at the NIH Clinical Center will undergo pre-injection, 24, 48 (optional) hours post-Ferumoxytol injection MRI consisting of T1 weighted (W), T2W and T2*W MRI at 3 Tesla magnet.
* In the dose finding cohorts, each dose (4mg/kg Fe, 6mg/kg Fe, 7.5mg/kg Fe) will have an equal number of patients (estimated enrollment will be 5 evaluable patients for each group, making a total of 3x5=15 patients) will be enrolled sequentially. In the lymph node involvement cohort, 5 evaluable subjects will be enrolled.
* Subjects in the dose finding cohorts will undergo clinically indicated prostatectomy, nodal dissection for prostate cancer; histology of resected lymph nodes will be correlated with imaging.
* Subjects in the lymph node involvement cohort may be scheduled to undergo prostatectomy and nodal dissection or core needle biopsy of the lymph node(s) as part of their clinical work-up and histology of resected or biopsied lymph nodes will be correlated with imaging.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subject must be male and be greater than or equal to 18 years old.
* Subject must have a histologically confirmed diagnosis of prostate cancer.
* Subjects enrolling in the lymph node involvement subgroup must have imaging evidence of lymph node involvement (with a size of greater than or equal to 1.5 cm).
* Subject must have Eastern Cooperative Oncology Group Performance score less than or equal to 2.

Subjects in the dose finding cohorts must be scheduled to undergo prostatectomy for presumed prostate cancer.

-Subjects must be scheduled to undergo prostatectomy for presumed prostate cancer

EXCLUSION CRITERIA:

* Subjects with known hypersensitivity and allergy to iron
* Subjects with evidence of iron overload with a pre-study ferritin level greater than 370 ng/ml and percent saturation of transferrin level greater than 40%. Patients with lab values above these limits may be included in the study if documented hematology consultation rules out hemochromatosis.
* Subjects with any coexisting medical or psychiatric condition that is likely to interfere with study procedures and/or results
* Subjects with severe claustrophobia unresponsive to oral anxiolytics
* Subjects with contraindications to MRI
* Subjects weighing >136 kg (weight limit for scanner table)
* Subjects with pacemakers, cerebral aneurysm clips, shrapnel injury, or other implanted electronic devices or metal not compatible with MRI.
* Subjects with abnormal liver function tests suggesting liver dysfunction (AST and ALT >2 times the upper limits of normal; total bilirubin, of >2 times the upper limits of normal or >3.0 mg/dl in patients with Gilbert s syndrome).
* Subjects with other medical conditions deemed by the principle investigator (or associates) or the sponsor to make the subject ineligible for protocol procedures.

INCLUSION OF WOMEN AND MINORITIES:

* Members of all races and ethnic groups are eligible for this trial.
* Women are excluded from this trial as prostate cancer does not occur in females.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-01-26; Primary Completion 2015-03-19 (Actual); Study Completion 2015-03-19 (Actual)

PRIMARY OUTCOMES:
Optimal dose of Ferumoxytol for enhancing lymph nodes | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Choyke, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Li W, Tutton S, Vu AT, Pierchala L, Li BS, Lewis JM, Prasad PV, Edelman RR. First-pass contrast-enhanced magnetic resonance angiography in humans using ferumoxytol, a novel ultrasmall superparamagnetic iron oxide (USPIO)-based blood pool agent. J Magn Reson Imaging. 2005 Jan;21(1):46-52. doi: 10.1002/jmri.20235. PMID 15611942
- [Background] Li W, Salanitri J, Tutton S, Dunkle EE, Schneider JR, Caprini JA, Pierchala LN, Jacobs PM, Edelman RR. Lower extremity deep venous thrombosis: evaluation with ferumoxytol-enhanced MR imaging and dual-contrast mechanism--preliminary experience. Radiology. 2007 Mar;242(3):873-81. doi: 10.1148/radiol.2423052101. PMID 17325072
- [Background] Neuwelt EA, Varallyay CG, Manninger S, Solymosi D, Haluska M, Hunt MA, Nesbit G, Stevens A, Jerosch-Herold M, Jacobs PM, Hoffman JM. The potential of ferumoxytol nanoparticle magnetic resonance imaging, perfusion, and angiography in central nervous system malignancy: a pilot study. Neurosurgery. 2007 Apr;60(4):601-11; discussion 611-2. doi: 10.1227/01.NEU.0000255350.71700.37. PMID 17415196